CLINICAL TRIAL: NCT03855891
Title: Evaluation of the Circulating Micro-RNA Profile Specificity in Patients With Different Stages of Atherosclerosis According to MSCT Coronary Angiography
Brief Title: Micro-RNA Profile in Patients With Different Stages of Atherosclerosis According to CTA
Acronym: CT-CA-miRNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Andrei N Rozhkov, MD, Post-graduate student of Department of of Preventive and Emergency Cardiology I.M. Sechenov First Moscow State Medical University, I.M. Sechenov First Moscow State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1741909-2019
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Ischemic Heart Disease; Atherosclerosis
Keywords: Ischemic Heart Disease; Atherosclerosis; micro-RNA; multislice spiral computed tomography; coronary angiography
MeSH Terms: conditions — Myocardial Ischemia; Atherosclerosis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): A group of patients with blood tests
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — Blood test for spectrum and level of cardiospecific micro-RNA

SUMMARY:
The main purpose of this single-center study is to determine the spectrum and levels of cardiospecific circulating microRNAs in patients with different stages of atherosclerosis according to 640-slice multispiral computed tomography (MSCT).

DETAILED DESCRIPTION:
The study will be conducted in two phases. Phase one. After signing the informed consent, patients with coronary heart disease, angina pectoris II-IV functional class, who underwent MSCT angiography of the coronary arteries for medical reasons, regulated in the relevant ESC and the Russian Society of Cardiology guidelines, will be included in the study. According to the results of MSCT, the participants will be divided into 4 groups: those with atherosclerotic plaques with signs of instability; those with stable atherosclerotic plaques without marked calcification; those with calcined atherosclerotic plaques; those with no signs of atherosclerosis of the coronary arteries. Plasma samples will be analyzed by microarray, using a cardiospecific set.

Phase two. Validation of the results obtained after the first phase will be performed on a larger sample of patients. Patients after signing an informed consent will also undergo MSCT angiography of coronary arteries and according to its results will be devided in 4 groups. To assess the level of microRNA expression in the blood of patients, real-time reverse transcription-polymerase chain reaction (RT-PCR) will be used.

The expected result of the study. For the first time ever, there will be determined the profile of circulating regulatory RNA in patients who underwent MSCT angiography of coronary arteries. Features of expression of circulating microRNAs will be compared with different severity degrees of the atherosclerotic process based on MSCT criteria. The results will be compared with each other (including the "control" group), which will allow to identify common patterns and specific differences.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient to participate in the study;
* Age 18-80;
* The presence of medical indications for MSCT angiography of coronary arteries in connection with suspected coronary heart disease.

Exclusion Criteria:

* Age less than 18 or more than 80;
* Pregnancy, breast-feeding;
* Patients who have not undergone (and do not plan) MSCT coronary angiography;
* Any surgical intervention on the heart in history;
* Severe heart failure (III-IV NYHA classes);
* History of myocardial infarction;
* The body mass index of 35 or more;
* More than twice the ALT and/or AST level;
* The presence of severe somatic pathology (except coronary atherosclerosis);
* Patient's refusal to participate in the study;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Determination of the profile of circulating microRNAs in patients with different degrees of severity of atherosclerotic process on the MSCT criteria basis. | 2 days
  Analysis of the spectrum and levels of cardiospecific circulating microRNAs in patients with different degrees of severity of atherosclerotic process on the MSCT criteria basis.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kopylov, Professor, Principal Investigator — Sechenov Univercity
Locations (1):
- IMSechenovMMA, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Data disclosure is not permitted by the local ethics committee. For more information about the study, you need to contact the principal investigator.